CLINICAL TRIAL: NCT07225725
Title: Community Health Support for Emergency Department-Presenting Head and Neck Cancer Patients: A Pilot to Improve Access to Timely Care
Brief Title: Access to Care Pilot for ED-Presenting Head and Neck Cancer Patients (ENRICH-HNC)
Acronym: ENRICH-HNC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Methodist University Hospital (Unknown); Regional One Health (Other); UTHSC Center for Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-10971-XP
Record Dates: First submitted 2025-11-04; First posted 2025-11-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Neoplasms; Emergency Department Presentation; Head and Neck Cancer (H&N)
Keywords: Emergency Department; Patient Navigation; Community Health Support; Health Equity; Cancer Care Access; Care Timeliness; Implementation Science; Engaging Navigators to Reduce Inequities in Cancer Health; ENRICH Program; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Emergencies

STUDY DESIGN:
Intervention Model Description: Single-arm, prospective feasibility pilot evaluating structured Community Health Support Specialist (CHSS) navigation initiated after emergency department discharge for adults presenting to the ED with suspected or newly diagnosed head and neck cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community Health Support Specialist (CHSS) Navigation (Experimental): Participants will receive structured, non-clinical navigation support from a trained Community Health Support Specialist (CHSS) initiated after emergency department discharge. CHSS outreach will occur by telephone or text message and will focus on identifying social and logistical barriers to timely cancer care (e.g., transportation, insurance, housing, communication), providing appropriate resource referrals, and reinforcing communication between patients and clinical care teams as needed. Each participant will receive a minimum of two CHSS contacts prior to initiation of definitive cancer treatment.
  Interventions: Behavioral: Community Health Support Specialist (CHSS) Navigation

INTERVENTIONS:
Behavioral: Community Health Support Specialist (CHSS) Navigation — This intervention consists of structured, non-clinical navigation delivered by trained Community Health Support Specialists (CHSS) as part of the Engaging Navigators to Reduce Inequities in Cancer Health (ENRICH) program. Following emergency department discharge and completion of electronic informed consent, CHSS staff conduct outreach by telephone or text message to identify and address social and logistical barriers to timely head and neck cancer care. Navigation activities may include assistance with transportation resources, insurance or financial navigation, connection to housing or community services, and reinforcement of communication between patients and clinical care teams. CHSS staff do not provide medical advice, schedule clinical appointments, or alter treatment plans. All navigation encounters are documented using standardized REDCap instruments.

SUMMARY:
Patients diagnosed with head and neck cancer (HNC) after presenting to an emergency department (ED) often face significant delays in diagnosis and treatment. These patients are frequently younger, underinsured, and experience multiple socioeconomic and systems-level barriers to accessing timely cancer care. Delays of more than 30 days have been associated with worse outcomes, including higher recurrence rates and reduced survival.

This pilot study will evaluate the feasibility and early impact of a community-based navigation program designed to improve access to timely care for ED-presenting HNC patients. The study embeds trained Community Health Support Specialists (CHSS) from the Engaging Navigators to Reduce Inequities in Cancer Health (ENRICH) program into the ED-to-treatment pathway. After ED discharge, CHSS staff will contact participants by telephone or text message to identify barriers to care-such as transportation, insurance, housing, or communication challenges-and connect them with appropriate community or institutional resources.

All participants will receive the CHSS navigation intervention. Outcomes will be compared with a historical cohort of similar ED-presenting HNC patients treated prior to program implementation. The primary outcomes are time from ED discharge to diagnostic biopsy and time from ED discharge to initiation of definitive treatment. Secondary outcomes include feasibility, measured as the proportion of participants who complete CHSS navigation, and exploratory analyses of the types of barriers identified and resolved.

Findings from this pilot will generate preliminary data to inform larger studies aimed at improving access, reducing disparities, and accelerating treatment for head and neck cancer patients who first present in the emergency setting.

DETAILED DESCRIPTION:
This is a single-arm, prospective pilot study evaluating the feasibility and process impact of embedding Community Health Support Specialist (CHSS) navigation within the emergency department (ED)-to-treatment pathway for patients with newly suspected or newly diagnosed head and neck cancer (HNC). The study will be conducted at two University of Tennessee Health Science Center (UTHSC)-affiliated hospitals: Methodist University Hospital and Regional One Health.

Eligible participants are adults aged 18 years or older who present to the ED with a new or suspected HNC involving the oral cavity, oropharynx, hypopharynx, larynx, salivary glands, skin, sinonasal region, nasopharynx, thyroid, or an unknown primary. Patients with prior established oncology care for HNC, those enrolled in hospice, incarcerated individuals, or patients who cannot be contacted by telephone will be excluded.

During routine clinical care in the ED, otolaryngology residents identify potentially eligible patients and introduce the study using an IRB-approved consent disclosure statement. ED activities are limited to screening and obtaining permission to contact; no informed consent or HIPAA authorization occurs in the ED.

After ED discharge, a trained study team member conducts the full informed consent process electronically using REDCap eConsent. Participants may review the consent form remotely with study staff and provide electronic signature with date/time acknowledgment. Only participants who complete electronic informed consent and HIPAA authorization are enrolled.

Following enrollment, CHSS specialists initiate outreach within 72 hours of ED discharge and provide structured, non-clinical navigation support through at least two telephone or text-based contacts prior to initiation of definitive cancer treatment. CHSS activities focus on identifying and addressing barriers to care, including transportation challenges, insurance or financial barriers, housing instability, and communication gaps. CHSS staff do not provide medical advice, schedule clinical appointments, or alter treatment plans. All encounters are documented using standardized REDCap case report forms.

The primary outcomes are (1) time from ED discharge to diagnostic biopsy and (2) time from ED discharge to initiation of definitive treatment. Secondary outcomes include feasibility, measured as the proportion of enrolled participants who complete CHSS navigation. Exploratory outcomes describe the types of social barriers identified, the proportion of barriers resolved, and patterns of navigation support.

Study data are entered and stored in REDCap, a secure, HIPAA-compliant database hosted by UTHSC. Outcomes for the pilot cohort will be compared with a historical control group of similar ED-presenting HNC patients treated at UTHSC-affiliated hospitals in the 24 months preceding program implementation. Analyses will use descriptive, non-parametric, and regression methods to estimate feasibility metrics and effect sizes to inform future multi-site studies.

This study is funded through the UTHSC Cancer Center's Access to Cancer Care Pilot Project and builds upon the Tennessee Department of Health-supported ENRICH program, which deploys CHSS specialists to reduce disparities in cancer care. Results will inform potential expansion of this navigation model to improve equity, timeliness, and outcomes for head and neck cancer patients presenting through the emergency department.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older
* Presentation to the emergency department (ED) with a new or suspected head and neck cancer (including oral cavity, oropharynx, hypopharynx, larynx, salivary gland, cutaneous, sinonasal, nasopharyngeal, thyroid, or metastatic disease with unknown primary)
* Residence within the regional catchment area of participating UTHSC-affiliated hospitals (Methodist University Hospital or Regional One Health)
* Ability to provide informed consent electronically using REDCap eConsent after ED discharge
* Has a valid telephone number for post-discharge contact

Exclusion Criteria

* Prior or ongoing established head and neck oncology care at the time of ED presentation
* Currently receiving hospice or palliative-only care
* Incarcerated individuals
* Inability to complete electronic informed consent (e.g., lack of decisional capacity or inability to complete consent even with staff assistance)
* Lacks reliable telephone access or is unable to be reached after three documented contact attempts by study staff
* Non-English or non-Spanish speaking when interpreter services are unavailable
* Expected survival less than four weeks, as determined by the treating clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Time From Emergency Department (ED) Presentation to Diagnostic Biopsy (Days) | Up to 90 days after ED discharge
  Interval (days) between the date of ED discharge from the index visit and the date of the first diagnostic biopsy procedure performed to evaluate suspected head and neck cancer.
Time From Emergency Department (ED) Presentation to Treatment Initiation (Days) | Up to 90 days after ED discharge
  Interval (days) between the date of ED discharge from the index visit and the start date of definitive treatment (surgery, radiation, systemic therapy, or combined modality) for head and neck cancer.

SECONDARY OUTCOMES:
Feasibility of Community Health Support Specialist (CHSS) Navigation | Up to 90 days after enrollment
  Proportion of enrolled participants who complete the CHSS navigation protocol, defined as documentation of at least two completed CHSS outreach contacts (telephone or text message) prior to initiation of definitive treatment or study completion.

OTHER OUTCOMES:
Number and Types of Social Barriers Identified During CHSS Encounters | Up to 90 days after enrollment
  Count and categorization of distinct social or logistical barriers (e.g., transportation, insurance, housing, communication) documented by CHSS staff across all encounters using standardized REDCap instruments.
Number of Barriers Resolved Through CHSS Intervention | Up to 90 days after enrollment
  Count of barriers documented as resolved by CHSS staff using standardized REDCap instruments. Resolution is defined as documentation that the participant was successfully linked to an appropriate resource/service or that the identified barrier was otherwise addressed.

CONTACTS AND LOCATIONS:
Overall Officials: David Schwartz, MD, Principal Investigator — University of Tennessee
Locations (2):
- United States (2):
  - Methodist University Hospital, Orlando, Florida
  - Regional One Health, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this is a small, minimal-risk feasibility study containing identifiable clinical data. Aggregate results may be shared in publications and presentations.

REFERENCES:
- See also: UTHSC news release describing the ENRICH program, a state-funded initiative led by Drs. Schwartz and Stewart to improve cancer care access through community health support specialists in West Tennessee. — https://news.uthsc.edu/uthsc-team-wins-2-75-million-from-state-to-improve-cancer-care-access-in-west-tennessee/
- See also: Official UTHSC Cancer Center webpage providing information about cancer research, pilot grant programs, and access-to-care initiatives supported by the institution. — https://uthsc.edu/cancer/